CLINICAL TRIAL: NCT01073761
Title: Pharmacokinetics of Darunavir/Ritonavir Once Daily and Atazanavir/Ritonavir Once Daily Over 72 Hours Following Drug Intake Cessation
Brief Title: Atazanavir/Ritonavir and Darunavir/Ritonavir PK Tail Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Dr Marta Boffito, St Stephen's AIDS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSAT 034
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: HIV; HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everybody (Experimental): All Subjects will receive the same intervention
  Interventions: Drug: darunavir/ritonavir then atazanavir/ritonavir

INTERVENTIONS:
Drug: darunavir/ritonavir then atazanavir/ritonavir — Phase 1: Oral darunavir/ritonavir 800/100 mg once daily for 10 days
  Phase 2: Oral atazanavir/ritonavir 300/100 mg once daily for 10 days
  Other Names: Prezista = TMC114; Norvir,; Reyataz = BMS-232632

SUMMARY:
The purpose of the study is to look at the levels of three HIV medications darunavir, ritonavir and atazanavir in the blood after the drug intake has been stopped in order to understand how long these drugs persist in blood for. The study will specifically look at these three drugs blood levels after taking them for 10 days everyday.

The main objective is to provide information on the potential safety (in terms of preventing virological failure and the development of resistance)of delaying drug doses occasionally by providing information on the decline in drug concentration after dosing has stopped.

DETAILED DESCRIPTION:
The long term use of and success of antiretroviral therapy (ART) is constrained by many factors including poor adherence and drug intolerance. Poor adherence (missing ART doses) may lead to the achievement of sub therapeutic drug plasma concentrations and virological failure. This could also be complicated by the development of resistance to ART which compromises future therapeutic options because of cross resistance within antiretroviral drug classes.

In medicine, successful adherence is supposed to mean taking at least 80% of doses. This is a concept, which has been inherited from the antihypertensive literature and anti-infective prescribing for therapeutic areas which from that of HIV prescribing in fundamental principles. The current absence of a curative therapy for HIV infection, means that in order to be effective, suppressive therapies need to be taken on an indefinite lifelong basis. The capacity for development of resistance of the virus means that successful adherence equates to a much higher rate of adherence than 80%. Moreover, in HIV therapy, successful adherence also means attention to a maximum interval between doses as well as dietary restriction at the time of dose intake.

Ideally, to guarantee long-term virological response, HIV-infected patients should take their ART every day at the same time. However, ART is for life and doses can be forgotten or delayed.

A recent survey confirmed the reasons why people miss their antiretroviral doses: they forget, they fall asleep, they are too busy, they are depressed, they are away from home, and their medicines make them sick (Mascolini www.thebody.com 2003).

Drug persistence (the presence of drug at a detectable level high enough to work) in plasma mainly depends on the half-life. Long half-life antiretroviral agents may allow for forgotten doses, if they are able to delay the decline of the drug level to sub-therapeutic concentrations for long enough for the patient to remember to take the drug. Boosted PI are characterized by different half lives, and therefore different abilities to persist in plasma.

Unfortunately, data on drug persistence in plasma are limited and whether drug doses can be forgotten and dosing delayed is unknown.

Therefore, the main objective of this study is to provide information on the potential safety (in terms of preventing virological failure and the development of resistance) of delaying drug doses occasionally by providing information on the decline in drug concentration after dosing has stopped.

Rationale for pharmacogenomic analysis

Pharmacogenetics holds promise in HIV treatment because of the complexity and potential toxicity of multi antiretroviral drug therapies that are prescribed for long periods. Thus far, few candidate genes have been examined for a limited number of allelic variants, but a number of confirmed associations have already emerged.

From a public health perspective, as antiretroviral medications become increasingly available to racially and ethnically diverse populations worldwide, understanding the genetic structures of each population may allow us to anticipate the impact of adverse responses, even in groups that were not represented in drug registration trials.

The existing literature on pharmacogenetic determinants of antiretroviral drug exposure, drug toxicity, as well as genetic markers associated with the rate of disease progression underline the recent advances which occurred in the past few years.

However, it is expected that larger-scale comprehensive genome approaches will profoundly change the landscape of knowledge in the future. Additional studies are needed to assess the implications for long-term responses to antiretroviral agents.

For this reason we plan to collect a single blood sample from each participant in our intensive pharmacokinetic studies, such as this one, in order to be able to investigate the association between genetic polymorphisms in drug disposition genes (such as those encoding for cytochrome P450 isoenzymes or transmembrane transporters) and drug exposure. A candidate gene approach will be utilised to examine loci of interest. This procedure will provide potentially important information on genetic influences on plasma drug concentrations and give insight into how to improve the management of HIV-infected patients by individualising therapy. These studies will not be powered for genetic associations but will enable us to build a data base of genotype-phenotype associations. Prospective genetic studies would need to be planned based on these preliminary data.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria within 28 days prior to the baseline visit:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements
2. Male or non-pregnant, non-lactating females
3. Between 18 to 65 years, inclusive
4. Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive.
5. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least one month after the study

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study.

1. Any significant acute or chronic medical illness
2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
3. Positive blood screen for hepatitis B surface antigen and/or C antibodies
4. Positive blood screen for HIV-1 and/or 2 antibodies
5. Current or recent (within 3 months) gastrointestinal disease
6. Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study
7. Exposure to any investigational drug or placebo within 3 months of first dose of study drug
8. Use of any other drugs (unless approved by the Investigator), including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug
9. Females of childbearing potential without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least 30 days after the end of the treatment period

19. Previous allergy to any of the constituents of the pharmaceuticals administered in this trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 30 days (excluding screening and follow-up)
  To assess the pharmacokinetics of darunavir/ritonavir once daily and atazanavir/ritonavir once daily over 72 hours following drug intake cessation

SECONDARY OUTCOMES:
Inter-Subject Variability | 30 days
  To assess the inter subject variability in darunavir and atazanavir plasma concentrations over 72 hours following drug intake cessation.
Safety and Tolerability | 30 day (excluding screening and follow up)
  To assess the safety and tolerability of darunavir/ritonavir and atazanavir/ritonavir over 10 days of administration
Pharmacogenetics | 30 day (excluding screening and follow up)
  To investigate the association between genetic polymorphisms in drug disposition genes and drug exposure

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Dr, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's Centre, London, United Kingdom